CLINICAL TRIAL: NCT00255814
Title: A Phase I Trial of Highly Conformal Radiation Therapy for Patients With Liver Metastases
Brief Title: Radiation Therapy in Treating Patients With Liver Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0438; CDR0000450766
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Metastatic Cancer
Keywords: liver metastases
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Radiation therapy dose level II: 4.0 Gy/fx (Other): Radiation therapy dose level II: 4.0 Gy/fraction
  Interventions: Radiation: radiation therapy
- Radiation therapy dose level III: 4.5 Gy/fx (Other): Radiation therapy dose level III: 4.5 Gy/fraction
  Interventions: Radiation: radiation therapy
- Radiation therapy dose level IV: 5.0 Gy/fx (Other): Radiation therapy dose level IV: 5.0 Gy/fraction
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This phase I trial is studying the side effects and best dose of radiation therapy in treating patients with liver metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of high dose per fraction, highly conformal radiotherapy in patients with liver metastases.

Secondary

* Determine the failure patterns and survival of patients treated with this regimen.
* Correlate dose-volume characteristics with possible toxic effects of this regimen in these patients.
* Determine the local control rate within irradiated fields in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study.

Patients undergo highly conformal radiotherapy (HCR) to the liver once daily, 5 days a week, for 2 weeks.

Cohorts of 6 patients receive escalating doses of HCR until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed periodically for 3 years.

PROJECTED ACCRUAL: A total of 18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Histologically confirmed non-lymphoma liver metastases
  * New radiographic liver lesions most consistent with metastases in a patient with known, histologically proven non-lymphoma cancer AND a previously negative CT scan, MRI, or PET/CT scan of the liver
* No more than 5 measurable lesions by contrast-enhanced liver CT scan, MRI, or PET/CT scan
* Liver metastases ≤ 8 cm
* Medically unfit for surgery OR lesions are surgically unresectable
* All intrahepatic disease must be encompassed within the study radiation field
* Extrahepatic disease outside the liver is allowed provided the hepatic disease is life-limiting
* At least 1,000 cc of normal liver
* No clinical ascites
* No CNS metastases

PATIENT CHARACTERISTICS:

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,800/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8 g/dL (transfusion allowed)

Hepatic

* No active hepatitis
* No clinically significant liver failure
* No underlying cirrhosis

Renal

* Not specified

Cardiovascular

* No congestive heart failure requiring hospitalization within the past 6 months
* No unstable angina pectoris requiring hospitalization within the past 6 months
* No transmural myocardial infarction within the past 6 months

Pulmonary

* No chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 3 years except non-melanomatous skin cancer or carcinoma in situ of the breast, oral cavity, cervix or primary liver metastasis
* No acute bacterial or fungal infection requiring IV antibiotics

PRIOR CONCURRENT THERAPY:

Chemotherapy

* At least 4 weeks since prior chemotherapy
* No concurrent chemotherapy
* No anthracyclines within 4 weeks after completion of study therapy (1 week for other chemotherapy)

Radiotherapy

* No prior radiotherapy to the region of study
* No concurrent intensity-modulated radiotherapy

Surgery

* Prior liver resection or ablative therapy allowed

Other

* No concurrent warfarin or IV heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-11; Primary Completion 2011-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To determine the maximally tolerated dose | From start of treatment to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Alan W. Katz, MD, Principal Investigator — James P. Wilmot Cancer Center; Laura A. Dawson, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (3):
- James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York, United States
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill Cancer Centre at McGill University, Montreal, Quebec